CLINICAL TRIAL: NCT02810639
Title: Pain Prevalence After Cesarean Section in Siriraj Hospital
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Sirilak Suksompong, Associate Professor, Mahidol University
Other Study IDs: 816/2554(EC3)
Record Dates: First submitted 2016-06-17; First posted 2016-06-23 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Pain, Postoperative
Keywords: pain
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Spinal morphine has been widely provided for acute postoperative analgesia. However, the analgesic effect of spinal morphine usually last 12-24 hours. Therefore the investigators are interested in the pain characteristics during the 2nd postoperative day. The investigators will also explore the regimens for pain therapy in our hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Cesarean section

Exclusion Criteria:

* History of drug addict

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing Cesarean section
Sampling Method: Non-Probability Sample
Enrollment: 297 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Number of patients who have moderate to severe pain after Cesarean section | 24-48 hours
  Number of patients who have moderate to severe pain after Cesarean section

CONTACTS AND LOCATIONS:
Overall Officials: Sirilak Suksompong, MD, Principal Investigator — Mahidol University
Locations (1):
- Sirilak Suksompong, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No